CLINICAL TRIAL: NCT02106897
Title: A Single-Ascending-Dose and Multiple-Ascending-Dose Study of BIIB059 in Healthy Volunteers and Subjects With Systemic Lupus Erythematosus
Brief Title: Study Evaluating the Safety, Tolerability, and Pharmacokinetics of Single Doses and Multiple Doses of BIIB059 (Litifilimab) in Healthy Volunteers and Participants With Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 230LE101; 2013-005361-39 (EudraCT Number)
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Systemic Lupus Erythematosus; Healthy Volunteers
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (19):
- Part 1, Cohort 1: BIIB059 0.05 mg/kg IV (Experimental): BIIB059 0.05 mg/kg IV dose, Once on Day 1
  Interventions: Drug: BIIB059 (litifilimab)
- Part 1, Cohort 2: BIIB059 0.3 mg/kg IV (Experimental): BIIB059 0.3 mg/kg IV dose, Once on Day 1
  Interventions: Drug: BIIB059 (litifilimab)
- Part 1, Cohort 3: BIIB059 1 mg/kg IV (Experimental): BIIB059 1 mg/kg IV dose, Once on Day 1
  Interventions: Drug: BIIB059 (litifilimab)
- Part 1, Cohort 4: BIIB059 3 mg/kg IV (Experimental): BIIB059 3 mg/kg IV dose, Once on Day 1
  Interventions: Drug: BIIB059 (litifilimab)
- Part 1, Cohort 5: BIIB059 10 mg/kg IV (Experimental): BIIB059 10 mg/kg IV dose, Once on Day 1
  Interventions: Drug: BIIB059 (litifilimab)
- Part 1, Cohort 6: BIIB059 20 mg/kg IV (Experimental): BIIB059 20 mg/kg IV dose, Once on Day 1
  Interventions: Drug: BIIB059 (litifilimab)
- Part 1, Cohort 7: BIIB059 50 mg SC (Experimental): BIIB059 50 mg SC dose, Once on Day 1
  Interventions: Drug: BIIB059 (litifilimab)
- Part 1, Cohort 1-6: Placebo IV (Placebo Comparator): Matching placebo IV dose, Once on Day 1
  Interventions: Drug: Placebo
- Part 1, Cohort 7: Placebo SC (Placebo Comparator): Matching placebo SC dose, Once on Day 1
  Interventions: Drug: Placebo
- Part 2, Cohort 8: BIIB059 20 mg/kg IV (Experimental): BIIB059 20 mg/kg IV dose, Once on Day 1
  Interventions: Drug: BIIB059 (litifilimab)
- Part 2, Cohort 8: Placebo IV (Placebo Comparator): Matching placebo IV dose, Once on Day 1
  Interventions: Drug: Placebo
- Part 3a, Cohort 9: BIIB059 20 mg SC (Experimental): BIIB059 20 mg SC dose, Every 4 weeks for 2 doses
  Interventions: Drug: BIIB059 (litifilimab)
- Part 3a, Cohort 10: BIIB059 50 mg SC (Experimental): BIIB059 50 mg SC dose, Every 4 weeks for 2 doses
  Interventions: Drug: BIIB059 (litifilimab)
- Part 3a, Cohort 11: BIIB059 150 mg SC (Experimental): BIIB059 150 mg SC dose, Every 4 weeks for 2 doses
  Interventions: Drug: BIIB059 (litifilimab)
- Part 3a, Cohort 12: BIIB059 300 mg or less SC (Experimental): BIIB059 300 mg or less SC dose, Every 2 weeks for 3 doses
  Interventions: Drug: BIIB059 (litifilimab)
- Part 3a, Cohort 9-12: Placebo SC (Placebo Comparator): Matching placebo SC dose, Every 4 weeks for 2 doses or every 2 weeks for 3 doses
  Interventions: Drug: Placebo
- Part 3b, Cohort 13: BIIB059 50 mg SC (Experimental): BIIB059 50 mg SC dose, Every 4 weeks for 2 doses
  Interventions: Drug: BIIB059 (litifilimab)
- Part 3b, Cohort 14: BIIB059 300 mg or less SC (Experimental): BIIB059 300 mg or less SC dose, Every 2 weeks for 3 doses
  Interventions: Drug: BIIB059 (litifilimab)
- Part 3b, Cohort 13-14: Placebo SC (Placebo Comparator): Matching placebo SC dose, Every 4 weeks for 2 doses or every 2 weeks for 3 doses
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIIB059 (litifilimab) — See Arm Descriptions
  Other Names: litifilimab
  Arms: Part 1, Cohort 1: BIIB059 0.05 mg/kg IV; Part 1, Cohort 2: BIIB059 0.3 mg/kg IV; Part 1, Cohort 3: BIIB059 1 mg/kg IV; Part 1, Cohort 4: BIIB059 3 mg/kg IV; Part 1, Cohort 5: BIIB059 10 mg/kg IV; Part 1, Cohort 6: BIIB059 20 mg/kg IV; Part 1, Cohort 7: BIIB059 50 mg SC; Part 2, Cohort 8: BIIB059 20 mg/kg IV; Part 3a, Cohort 10: BIIB059 50 mg SC; Part 3a, Cohort 11: BIIB059 150 mg SC; Part 3a, Cohort 12: BIIB059 300 mg or less SC; Part 3a, Cohort 9: BIIB059 20 mg SC; Part 3b, Cohort 13: BIIB059 50 mg SC; Part 3b, Cohort 14: BIIB059 300 mg or less SC
Drug: Placebo — See Arm Descriptions
  Arms: Part 1, Cohort 1-6: Placebo IV; Part 1, Cohort 7: Placebo SC; Part 2, Cohort 8: Placebo IV; Part 3a, Cohort 9-12: Placebo SC; Part 3b, Cohort 13-14: Placebo SC

SUMMARY:
The primary objective of Parts 1 and 2 is to evaluate the safety and tolerability of either single-ascending intravenous (IV) doses or a single subcutaneous (SC) dose of BIIB059 (litifilimab) in healthy volunteers (HV), and a single IV dose in participants with Systemic Lupus Erythematosus (SLE). The primary objective of Part 3 is to evaluate the safety and tolerability of multiple SC doses of BIIB059 in healthy volunteers and in participants with SLE.

Secondary objectives of Parts 1 and 2 are as follows: To estimate the PK parameters of single-ascending IV doses of BIIB059 in healthy volunteers and a single IV dose of BIIB059 in participants with SLE; To estimate the PK parameters and bioavailability (F) of a single SC dose of BIIB059 in healthy volunteers; To evaluate the immunogenicity of BIIB059 administered to healthy volunteers and participants with SLE. Secondary objectives of Part 3 are as follows: To estimate the PK parameters of multiple SC doses of BIIB059 in healthy volunteers and in participants with SLE; To evaluate the immunogenicity of BIIB059 administered SC to healthy volunteers and participants with SLE.

DETAILED DESCRIPTION:
Part 1 (single ascending dose in healthy volunteers) has closed to enrollment.

ELIGIBILITY:
Part 1: Key Inclusion Criteria For Healthy Volunteers:

* Be in good health as determined by the Investigator, based on medical history, physical examination, and 12-lead ECG.
* Body mass index (BMI) between 18 and 30 kg/m2 and body weight ≥45 kg.

Part 1: Key Exclusion Criteria For Healthy Volunteers:

* History of or positive test results at screening for the following: for human immunodeficiency virus (HIV), hepatitis C virus antibody (HCV Ab), hepatitis B virus (defined as positive for hepatitis B surface antigen [HBsAg] or hepatitis B core antibody [HBcAb]).
* - History of chronic, recurrent, or recent serious infection (e.g., pneumonia, septicemia) as determined by the Investigator within 3 months prior to screening and randomization.
* History of severe allergic or anaphylactic reactions or history of allergic reactions likely to be exacerbated by any component of the study drug.
* History of any clinically significant cardiovascular, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, or other major disease, as determined by the Investigator.
* Any live or attenuated immunization/vaccination within 1 month prior to randomization or planned to occur during the study period.
* Blood donation (1 unit or more) within 1 month prior to randomization.
* Vigorous exercise (e.g., jogging, swimming laps, heavy gardening, hiking uphill, etc.) within 48 hours prior to Day -1

Part II: Key Inclusion Criteria for SLE Participants:

* Definite SLE for at least 6 months duration or anti-dsDNA antibody, prior to screening.
* Presence of active lupus skin disease including acute, sub acute, and/or chronic cutaneous lupus (e.g., discoid) at the time of screening and randomization.
* BMI between 18 and <40 kg/m2 and body weight ≥45 kg.

Part II: Key Exclusion Criteria for SLE Participants:

* Active neuropsychiatric SLE including but not limited to the following: seizure, new or worsening impaired level of consciousness, psychosis, delirium or confusional state, aseptic meningitis, ascending or transverse myelitis, chorea, cerebellar ataxia, mononeuritis multiplex, or demyelinating syndromes.
* History of chronic, recurrent, or recent serious infection (e.g., pneumonia, septicemia) as determined by the Investigator within 3 months prior to screening and randomization.
* Symptoms of bacterial or viral infection (including upper respiratory tract infection) within 28 days prior to randomization.
* History of severe allergic or anaphylactic reactions or history of allergic reactions likely to be exacerbated by any component of the study drug.
* Evidence of skin conditions other than lupus skin disease (e.g., eczema) at screening or at the time of randomization that would interfere with evaluations of the effect of study treatment on lupus skin disease.
* Treatment with oral prednisone >15 mg daily (or equivalent). Any prednisone regimen must be stable for at least 28 days before randomization and expected to remain stable for the duration of the study.
* Treatment with any antibiotics within 14 days prior to randomization.

Part IIIa: Key Inclusion Criteria for Healthy Volunteers :

* Must be in good health as determined by the Investigator, based on medical history, physical examination, and 12-lead ECG.
* Must have a body mass index (BMI) between 18 and 30 kg/m2 and body weight ≥45 kg.

Part IIIa: Key Exclusion Criteria for Healthy Volunteers:

* History of chronic, recurrent, or recent serious infection (e.g., pneumonia, septicemia) as determined by the Investigator within 3 months prior to screening and randomization
* History of severe allergic or anaphylactic reactions or history of allergic reactions likely to be exacerbated by any component of the study treatment.
* Treatment with any antibiotics within 14 days prior to randomization.

Part IIIb: Key Inclusion Criteria for SLE Participants:

* Definite SLE for at least 6 months duration prior to screening
* Presence of active lupus skin disease including acute, subacute, and/or chronic cutaneous lupus (e.g., discoid), and/or hypocomplementemia , and/or positive anti-dsDNA antibody at the time of screening.
* Must have a BMI between 18 and <40 kg/m2 and body weight ≥45 kg.

Part IIIb: Key Exclusion Criteria for SLE Participants:

* Active neuropsychiatric SLE including but not limited to the following: seizure, new or worsening impaired level of consciousness, psychosis, delirium or confusional state, aseptic meningitis, ascending or transverse myelitis, chorea, cerebellar ataxia, mononeuritis multiplex, or demyelinating syndromes.
* History of chronic, recurrent, or recent serious infection (e.g., pneumonia, septicemia) as determined by the Investigator within 3 months prior to screening and randomization.
* History of severe allergic or anaphylactic reactions or history of allergic reactions likely to be exacerbated by any component of the study drug.
* Treatment with any antibiotics within 14 days prior to randomization.

NOTE: Other protocol-defined inclusion/exclusion Criteria May Apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2014-04-30 (Actual); Primary Completion 2016-05-24 (Actual); Study Completion 2016-05-24 (Actual)

PRIMARY OUTCOMES:
Number of Participants that Experience Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to Week 32

SECONDARY OUTCOMES:
Area Under the Concentration-Time Curve from Time 0 Extrapolated to Infinity (AUCinf) of BIIB059 | Up to Week 32
Maximum Observed Concentration (Cmax) of BIIB059 | Up to Week 32
Time to Reach Maximum Observed Concentration (Tmax) of BIIB059 | Up to Week 32
Terminal Elimination Half-Life (t1/2) of BIIB059 | Up to Week 32
Clearance (CL) of BIIB059 | Up to Week 32
Apparent Clearance (CL/F) of BIIB059 | Up to Week 32
  For SC cohorts only
Volume of Distribution (Vss) of BIIB059 | Up to Week 32
Apparent Volume of Distribution (Vz/F) of BIIB059 | Up to Week 32
  For SC cohorts only
Bioavailability (F) for a single SC dose of BIIB059 | Up to Week 32
Absorption Rate Profile for a Single SC Dose of BIIB059 | Up to Week 32
Number of Participants Who Develop Serum Anti-BIIB059 Antibodies | Up to Week 32

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (5):
- United States (5):
  - Research Site, Anniston, Alabama
  - Research Site, Birmingham, Alabama
  - Research Site, Orlando, Florida
  - Research Site, Great Neck, New York
  - Research Site, Duncansville, Pennsylvania

REFERENCES:
- [Derived] Furie R, Werth VP, Merola JF, Stevenson L, Reynolds TL, Naik H, Wang W, Christmann R, Gardet A, Pellerin A, Hamann S, Auluck P, Barbey C, Gulati P, Rabah D, Franchimont N. Monoclonal antibody targeting BDCA2 ameliorates skin lesions in systemic lupus erythematosus. J Clin Invest. 2019 Mar 1;129(3):1359-1371. doi: 10.1172/JCI124466. Epub 2019 Feb 18. PMID 30645203